CLINICAL TRIAL: NCT00295256
Title: Randomized Trial to Evaluate the Effectiveness of Nurse Case Management on High-Risk Pregnancy Outcomes
Brief Title: Randomized Trial to Evaluate the Effectiveness of Nurse Case Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M630-430-2029; IRB number 05-01-28-03
Record Dates: First submitted 2006-02-22; First posted 2006-02-23 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes; Gestational Diabetes; Hypertension; Preterm Delivery
Keywords: randomized trial; diabetes; pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational; Hypertension; Premature Birth; Diabetes Mellitus

INTERVENTIONS:
Behavioral: nurse case manager

SUMMARY:
The management of high-risk pregnancies require substantial use of medical resources. Our goal is to determine the effectiveness of a nurse case management program in which case managers are assigned to patients with high-risk conditions.

Our hypothesis is that women with diabetes in pregnancy or hypertension who are assigned a nurse case manager will have lower glucose levels and lower blood pressure levels

DETAILED DESCRIPTION:
We will recruit 50 women for each arm of the study. We we conduct a stratified randomization (by disease) in which women are randomized to a nurse case manager who provides on-going face-to-face contact compared to women who are assigned to a case manager with telephone contact only.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, gestational diabetes, preterm labor, hypertensive disease

Exclusion Criteria:

* No telephone; ability to provide consent; english-speaking

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Outcomes measures are mean fasting glucose levels, mean systolic pressure and mean diastolic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Nicholson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States